CLINICAL TRIAL: NCT02328261
Title: Icotinib in Treating Patients With Advanced Nasopharyngeal Carcinoma: A Phase II, Multi-center, Open-label Study
Brief Title: A Phase II Study of Icotinib in Treating Patients With Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV21
Record Dates: First submitted 2014-11-24; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Icotinib (Experimental): Icotinib (125 mg tablet) is orally administered three times daily
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Icotinib (125 mg tablet) is orally administered three times daily until disease progression or unaccepted toxicity.
  Other Names: Conmana

SUMMARY:
This is a phase 2 study to evaluate the efficacy of single-agent icotinib in patients with advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This phase 2 study is aimed to evaluate the efficacy of single-agent icotinib in patients with pretreated, advanced nasopharyngeal carcinoma. The primary endpoint is disease control rate (DCR).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced NPC
* Patients must be platinum-resistant defined as recurrence or progression of disease <6 months since previous treatment with a platinum based treatment regimen.
* Measurable disease per RECIST
* Adequate organ and marrow function
* Capable of understanding and complying with the protocol, and written informed consent

Exclusion Criteria:

* Prior treatment with gefitinib, erlotinib, or other drugs that target EGFR
* Patients must not be receiving any other investigational agents
* Other serious illness or medical condition including unstable cardiac disease requiring treatment, history of significant neurologic or psychiatric disorders (including psychotic disorders, dementia, or seizures), or active uncontrolled infection
* Women who are pregnant or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Disease control rate(DCR) | At least 8 weeks

SECONDARY OUTCOMES:
Progression-free survival | At least 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Hu, MD, Principal Investigator — The first affliated hospital of Guangxi medical university